CLINICAL TRIAL: NCT03628391
Title: Efficacy of Haloperidol to Decrease the Burden of Delirium in Adult Critically Ill Patients (EuRIDICE): a Prospective Randomised Multi-center Double-blind Placebo-controlled Clinical Trial
Brief Title: Haloperidol for Delirium in Adult Critically Ill Patients
Acronym: EuRIDICE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped because of futility of being able to reach a one-day difference between treatment groups in the primary outcome of DCFD in the intended sample size.
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Mathieu van der Jagt, Principal Investigator / Medical Doctor, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC-2017-115/NL62689.078.17
Record Dates: First submitted 2017-10-09; First posted 2018-08-14 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Delirium; Critical Illness; Intensive Care Psychosis; Cognitive Impairment; Cognitive Decline
Keywords: delirium; intensive care unit; critical illness; cognitive impairment
MeSH Terms: conditions — Delirium; Critical Illness; Cognitive Dysfunction | interventions — Haloperidol

STUDY DESIGN:
Intervention Model Description: Randomised controlled double-blind placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo and haloperidol (verum) will have the same appearance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- haloperidol (Active Comparator): study drug will be titrated based on delirium, diagnosed with a validated screening instrument (CAM-ICU or ICDSC), starting with 2.5mg IV q8h and titrated to a maximum of 5mg IV q8h.
  Agitation and hallucinations will be managed according to a pre-specified protocol in both treatment arms. First the study drug will be increased when agitation or delirium remain present. Further options include mainly the use of alfa-2 agonists (agitation) or atypical antipsychotic drugs (hallucinations).
  Interventions: Drug: Haloperidol
- placebo (Placebo Comparator): study drug will be titrated based on delirium, diagnosed with a validated screening instrument (CAM-ICU or ICDSC), starting with 2.5mg IV q8h and titrated to a maximum of 5mg IV q8h.
  Agitation and hallucinations will be managed according to a pre-specified protocol in both treatment arms. First the study drug will be increased when agitation or delirium remain present. Further options include mainly the use of alfa-2 agonists (agitation) or atypical antipsychotic drugs (hallucinations).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — haloperidol for ICU delirium, titrated on validated screening tool-based diagnosis
  Other Names: not any
  Arms: haloperidol
Drug: Placebo — placebo for ICU delirium, titrated on validated screening tool-based diagnosis
  Arms: placebo

SUMMARY:
The EuRIDICE trial will study whether haloperidol as a first line treatment for ICU delirium reduces delirium duration (and severity). Adverse outcomes typically associated with delirium will also be studied and include long term cognition, functional outcome and quality of life. Further, patient and family experiences and cost-effectiveness will be assessed. Finally, safety concerns associated with the use of haloperidol in this vulnerable population will be studied.

DETAILED DESCRIPTION:
BACKGROUND. Although widely used, the efficacy and safety of haloperidol for delirium in critically ill adults remain unclear. A randomised controlled trial is warranted to study the effect of haloperidol on delirium or coma, long-term outcomes, safety concerns, and cost-effectiveness.

SUMMARY.

The investigators will perform a multi-center, randomised, double-blind, placebo-controlled clinical trial to evaluate the use of haloperidol for delirium treatment in 742 critically ill adults with delirium. Days spent without delirium- or coma in the first 14 days after randomisation is the primary outcome. Study drug will be initiated at 2.5mg IV q8h and increased after 24 hours to 5mg IV q8h if delirium persists. Study drug dose will be tapered when delirium has resolved during 24 hours. All patients will be managed with a standardized pain, agitation and delirium protocol. Standard operating procedures for agitation (analgesia titration, alpha2 agonists) and hallucination management (atypical antipsychotics) will be implemented to accommodate possible imbalances of these symptoms in both treatment arms. Open-label haloperidol administration is discouraged during the trial. The sample size provides a power of 90% to detect statistically significant results (p<.05) and a true treatment difference of one day for the primary outcome between trial arms.

This trial is expected to answer the clinically relevant question whether haloperidol still deserves a place in ICU delirium management. The primary outcome (delirium- and coma-free days) will be related to the secondary outcomes cognitive dysfunction, functional and psychological outcomes and patient- and family experiences. An extensive cost-effectiveness analysis will be done. Mortality at one year and safety concerns of haloperidol (QTc prolongation on EKG and rigidity) will be assessed as secondary endpoints. In conclusion, this large multicentre trial will assess efficacy and safety of haloperidol for ICU delirium.

ELIGIBILITY:
Inclusion Criteria for randomisation:

1. Delirium, as assessed with the Intensive Care Delirium Screening Checklist - ICDSC: ≥4 or Confusion Assessment Method for the ICU - CAM-ICU: positive). NB Delirium can occur in the course of ICU admission or be present at admission.
2. Written Informed Consent is obtained from patient or legal representative
3. Complies with inclusion criteria but NOT exclusion criteria for eligibility:

Eligibility

Inclusion criteria for eligibility

1. Age ≥ 18 years
2. Admitted to ICU.

Exclusion criteria for eligibility

1. Admitted to ICU with a neurological diagnosis (such as acute stroke, traumatic brain injury, intracranial malignancy, anoxic coma). Previous non-acute stroke or other previous neurological condition without cognitive deterioration is not an exclusion criterion.
2. Pregnancy (to be excluded by pregnancy test in women of child baring age)
3. History of ventricular arrhythmia including "torsade de pointes" (TdP)
4. Known allergy to haloperidol
5. History of dementia or an Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score ≥ 4
6. History of malignant neuroleptic syndrome or parkinsonism (either Parkinson's disease or another hypokinetic rigid syndrome)
7. Schizophrenia or other psychotic disorder
8. Inability to conduct valid delirium screening assessment (e.g. coma, deaf, blind) or inability to speak Dutch
9. The patient is expected to die within 24 hours, or is expected to leave the ICU within 24 hours after evaluation (may be reassessed daily)

Exclusion Criteria for randomisation:

1. Prolonged QT-interval (QTc > 500ms)
2. (recent) "torsade de pointes" (TdP)
3. (recent) malignant neuroleptic syndrome or parkinsonism
4. Evidence of acute alcohol (or substance) withdrawal requiring pharmacological intervention (e.g. benzodiazepines or alfa-2 agonist) to treat
5. IQCODE not assessed
6. The patient is expected to die within 24 hours, or is expected to leave the ICU within 24 hours.
7. No (previously) signed informed consent by patient or representative
8. Current participation in another intervention trial that is evaluating a medication, device or behavioural intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
delirium- and coma-free days | within the first 14 days after randomisation
  days without brain dysfunction (=delirium OR coma) while at the ICU

SECONDARY OUTCOMES:
Cognitive deterioration: Global cognitive functioning | 3 and 12 months
  Global cognitive functioning as assessed with the Montreal Cognitive Assessment (MOCA). Total score will be reported, with a range of 0-30 (higher values representing better cognitive functioning).
Cognitive deterioration: Verbal learning and memory | 3 and 12 months
  Auditory-verbal learning and memory will be assessed with the Rey Auditory Verbal Learning Test. Three subscores will be reported: total correct words in 5 trials (range: 0 -75), total correct words after delay (range: 0-15) and total correct words at recognition (range: 0-30).
Cognitive deterioration: Semantic fluency | 3 and 12 months
  Semantic fluency will be tested with the Semantic Category Fluency Test. The amount of animals given within a time of 60 seconds will represent the score.
Cognitive deterioration: Working memory | 3 and 12 months
  Working memory will be assessed using the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III). Subscales will be reported for both digit span under forward and backward recall conditions. In addition, a total score will be reported, which equals the sum of both separate digit spans.
Cognitive deterioration: Cognitive flexibility | 3 and 12 months
  Cognitive flexibility, one of the executive funcions, will be assessed with the Trialmaking tests A and B. The total amount of seconds needed to finish each test will be reported, with less seconds needed representing better cognitive flexibility.
Cognitive deterioration: Word retrieval | 3 and 12 months
  Word retrieval is tested with the Boston Naming Test (30-item version). The total score (range: 0-30) represents the amount of correct answered drawings.
Anxiety and depression | 3 and 12 months
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS). Two subscales will be reported, one for anxiety symptoms (range: 0-21) and one for depression symptoms (range: 0-21). Higher values represent a worse outcome. A subscore >8 indicates anxiety or depression, respectively.
Functional outcome | 3 and 12 months
  Health-related quality of life will be assessed with the Short Form-35 (SF-36). Nine subscales will be reported on a 0 - 100 scale: physical functioning, role functioning - physical, bodily pain, general health, vitality, social functioning, role functioning - emotional, mental health and reported health transition. Higher values represent a better health-related quality of life.
mortality | 28 days and 1 year
  mortality
length of stay at ICU | days of ICU stay (time in days from ICU admission until ICU discharge). Assessed up to a maximum of 12 months after randomisation (end of follow-up period).
  length of stay at ICU (days)
Adverse drug associated events: prolonged QTc by EKG | while on study drug treatment during study period at ICU (up to 14 days after randomisation)
  prolonged QTc by EKG (ms)
Adverse drug associated events: muscle rigidity and other associated movements disorders | while on study drug treatment during study period at ICU (up to 14 days after randomisation)
  muscle rigidity and other associated movements disorders [measured with the Simpson Angus Scale]
Adverse drug associated events: ventricular arrhythmia's | during study period at ICU (up to 14 days after randomisation)
  ventricular arrhythmia's including torsade de pointes
Patients' memories related to their ICU stay | at discharge from hospital (up to a maximum of 12 months after randomisation = end of follow-up period) and 3 months after randomisation
  Patients' memories for their ICU stay will be evaluated with the ICU Memory Tool (ICU-MT). Subscores will be reported for factual memories (range: 0-11), delusion memories (range: 0-6) and memories of feelings (range: 0-4).
Patients' and family-members' experiences related to delirium | at discharge from hospital (up to a maximum of 12 months after randomisation = end of follow-up period) and 3 months after randomisation
  Delirium recall and distress related to the delirium episode will be assessed with the Delirium Experience Questionnaire (DEQ). Scores will represent whether patients remember their delirium episode. In addition, a score representing delirium-related distress levels (range: 0-4, with higher values representing more distress) will be reported for both patients and family-members.
Caregiver Strain | at 3 months after randomisation
  The strain experienced by family-members or relatives will be assessed with the Caregiver Strain Index. A total score (range: 0-13) will be reported, with higher values representing higher experienced strain.
Posttraumatic stress syndrome | at 3 months after randomisation
  Posttraumatic stress symptoms in patients and families will be assessed with the Impact of Event Scale - Revised (IES-R). A mean total IES-R score will be reported (range: 0-4), with posttraumatic stress disorder defined as a mean IES-R score ≥ 1.6. In addition, subscores will be reported for intrusion, avoidance and hyperarousal (range: 0-4).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu van der Jagt, MD PhD, Principal Investigator — Erasmus University Medical Center Rotterdam, The Netherlands
Locations (8):
- Netherlands (8):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - IJsselland Hospital, Capelle aan den IJssel
  - Albert Schweitzer Hospital, Dordrecht
  - Radboudumc, Nijmegen
  - ErasmusMC, Rotterdam
  - Franciscus Gasthuis (Hospital), Rotterdam
  - Ikazia Hospital, Rotterdam
  - Maasstad Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided
Can be retrieved after contacting the principal investigator

REFERENCES:
- [Derived] Smit L, Slooter AJC, Devlin JW, Trogrlic Z, Hunfeld NGM, Osse RJ, Ponssen HH, Brouwers AJBW, Schoonderbeek JF, Simons KS, van den Boogaard M, Lens JA, Boer DP, Gommers DAMPJ, Rietdijk WJR, van der Jagt M; EuRIDICE study group. Efficacy of haloperidol to decrease the burden of delirium in adult critically ill patients: the EuRIDICE randomized clinical trial. Crit Care. 2023 Oct 30;27(1):413. doi: 10.1186/s13054-023-04692-3. PMID 37904241
- [Derived] Smit L, Trogrlic Z, Devlin JW, Osse RJ, Ponssen HH, Slooter AJC, Hunfeld NGM, Rietdijk WJR, Gommers D, van der Jagt M; EuRIDICE study group. Efficacy of halopeRIdol to decrease the burden of Delirium In adult Critically ill patiEnts (EuRIDICE): study protocol for a prospective randomised multi-centre double-blind placebo-controlled clinical trial in the Netherlands. BMJ Open. 2020 Sep 23;10(9):e036735. doi: 10.1136/bmjopen-2019-036735. PMID 32967873